CLINICAL TRIAL: NCT06044324
Title: A Prospective Study on the Efficacy and Safety of Transcranial Magnetic Stimulation Intervention for Treatment-Resistant Depression Guided by Positron Emission Tomography Imaging
Brief Title: Positron Emission Tomography in Transcranial Magnetic Stimulation Intervention for Treatment-resistant Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20240155C-R1
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Treatment Resistant Depression; Visual Perceptual Weakness
Keywords: Repetitive Transcranial Magnetic Stimulation; PET/MRI
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation (Active Comparator): Stimulation site: According to the localization of neural orientation navigation system, magnetic resonance data was read in Brainsight software, and three-dimensional brain reconstruction was carried out. The stimulation target was located in the coordinates of Montreal Neurological Institute (MNI), which was located in the left middle temporal (-43, -73, 10). Treatment intensity was 100% exercise threshold, continuous 10Hz stimulation, repeated 75 times, that is, 3000 pulses per treatment, 2 times a day, stimulation lasted for 4 seconds with a 26-second interval for 37.5 minutes, continuous stimulation for 5 days, 2 days rest interval, and 5 days of continuous stimulation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- HC observation (No Intervention): Collect data on healthy controls without stimulation. The subjects get clinical evaluation, blood sample collection, positron emission tomography-magnetic resonance scanning, and electrophysiological monitoring.

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Participants in the active stimulation group will receive the high frequency rTMS to left middle temporal visual area. The left middle temporal visual area will be targeted utilizing the neuronavigation system. Stimulation intensity will be standardized at 100% of RMT.
  Stimulation will be delivered to the left middle temporal visual area using an NTK-TMS-II100 TMS device,is compatible with the Brainsight TMS navigation system.
  Arms: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Major depressive disorder (MDD) exhibit reduced visual motor perception, which affects prognosis. Metabolic substance changes and abnormal neural activity in the middle temporal visual area (MT) mediate this perceptual dysfunction. The main questions are: •there is no conclusive evidence of impairment of visual motion suppression in treatment-resistant depression (TRD); •it is unknown that functional abnormalities in the MT of TRD patients mediate possible changes in visual perception •lack of treatment for deficit in visual motor perception; •mechanisms behind the intervention process need to be explored. The goal of this clinical trial is to understand the function of visual motor perception in TRD, to validate the effect of the MT on visual motion perception and to explore the effectiveness of the intervention as well as the neurophysiological mechanisms.

This study was planned to •explore any differences in visual motor perception and function of MT between TRD and healthy controls; •analyze the influence of neurobiological changes in MT and related brain regions on visual motion perception; •investigate the effects of rTMS intervention in MT for treatment of impaired visual perception function in TRD; •studying potential therapeutic mechanisms by PET/MRI imaging.

Participants will divide into TRD group and HC group. Clinical symptoms, scales, visual perception suppression index, PET/MRI, electrophysiology and other clinical data were collected at baseline for both two groups. TRD group received high-frequency rTMS stimulation targeting the MT. Besides, psychological scales, visual suppression index, PET/MRI, electrophysiology and other clinical data were collected during the intervention and after treatment.

The researchers will •compare the differences in visual perceptual function and neurobiological characteristics between the TRD group and the HC group in baseline; •analyze the impact of MT and related brain regions in visual motion perception; •compare the suppression index before and after intervention in TRD to discuss the feasibility of rTMS stimulation targeting the MT to improve visual motion perception abnormalities；•utilize the changes in clinical data of PET/MRI and electrophysiology before and after the treatment of TRD group to explore the possible underlying mechanisms during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

1. Receive two or more adequate doses and courses of antidepressant drugs in different mechanisms that were not effective and had been stable for more than 6 weeks on antidepressant medication prior to enrollment, with non-responsiveness defined as a decrease in HAMD-24 score of <50%.
2. 24-item Hamilton Depression Scale (HAMD-24) ≥ 20.
3. Normal or corrected to normal vision.
4. Ability to complete spatial suppression psychophysical experiment.
5. education background above the college degree.
6. Age 18-45 years, regardless of gender.
7. Right-handedness.
8. Han Chinese.
9. Signed a written informed consent, willing to participate in the study and be evaluated.

Exclusion Criteria:

1. Co-morbid other mental disorders, including: schizophrenia, mental retardation, substance dependence, etc.
2. Patients with metal objects in the body or with other contraindications to PET-MRI scanning
3. Patients with severe or unstable somatic diseases
4. Women during pregnancy or lactation, and women of childbearing age with positive urine HCG test results during the screening period
5. Benzodiazepines were taken during the experimental period
6. Other conditions that, in the opinion of the investigator, exist that make participation in this clinical trial inappropriate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Suppression Index after treatment | Baseline
  Suppression Index (SI) defined as the difference of log10 thresholds for large versus small stimuli of gratings, is able to quantify the suppression strength. The higher the numerical value, the more severe the visual motor perception deficit.
Change in Suppression Index after treatment | 2 weeks
  Suppression Index (SI) defined as the difference of log10 thresholds for large versus small stimuli of gratings, is able to quantify the suppression strength. The higher the numerical value, the more severe the visual motor perception deficit.
Hamilton Depression Scale (24-items) Total Score Change | Baseline
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. The higher scores representing more severe levels of depression. Remission is defined as HAM-D24 ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.
Hamilton Depression Scale (24-items) Total Score Change | 2 weeks
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. The higher scores representing more severe levels of depression. Remission is defined as HAM-D24 ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.
Change in synaptic density using positron emission tomography/magnetic resonance imaging | Baseline
  Positron emission tomography/magnetic resonance imaging (PET/MRI) is a fusion of PET and MRI, which integrates pathophysiological changes with morphological structure. Research using PET/MRI in major depression has shown that there are alterations in the snyaptic density of certain brain regions in people with the condition and synaptic dysfunction in the dorsolateral prefrontal cortex may have implications for the downstream organization of functional networks. The SV2A radioligand [11C]UCB-H can examine snyaptic density in human brain. And brain structure, function connectivity and spectrum of metabolic substances can be measured by MRI. Overall, PET/MRI has advantages for the diagnosis of major depression and the evaluation of treatment effects.
Change in synaptic density using positron emission tomography/magnetic resonance imaging | 2 weeks
  Positron emission tomography/magnetic resonance imaging (PET/MRI) is a fusion of PET and MRI, which integrates pathophysiological changes with morphological structure. Research using PET/MRI in major depression has shown that there are alterations in the snyaptic density of certain brain regions in people with the condition and synaptic dysfunction in the dorsolateral prefrontal cortex may have implications for the downstream organization of functional networks. The SV2A radioligand [11C]UCB-H can examine snyaptic density in human brain. And brain structure, function connectivity and spectrum of metabolic substances can be measured by MRI. Overall, PET/MRI has advantages for the diagnosis of major depression and the evaluation of treatment effects.

SECONDARY OUTCOMES:
Change in Suppression Index after treatment | 1 week
  Suppression Index (SI) defined as the difference of log10 thresholds for large versus small stimuli of gratings, is able to quantify the suppression strength. The higher the numerical value, the more severe the visual motor perception deficit.
Change in Suppression Index after treatment | 6 weeks
  Suppression Index (SI) defined as the difference of log10 thresholds for large versus small stimuli of gratings, is able to quantify the suppression strength. The higher the numerical value, the more severe the visual motor perception deficit.
Change in the score of Visual Analog Scale (VAS) | Baseline
  Subjective experience of time was measured by the VAS, which consists of a 100-mm vertical line representing the experience of time from slowest (i.e., -50 mm) to fastest (i.e., +50 mm). In this nonverbal dimensional task, subjects were asked to label how fast or slow they experienced the flow of time on the day of the survey.
Change in the score of Visual Analog Scale (VAS) | 1 week
  Subjective experience of time was measured by the VAS, which consists of a 100-mm vertical line representing the experience of time from slowest (i.e., -50 mm) to fastest (i.e., +50 mm). In this nonverbal dimensional task, subjects were asked to label how fast or slow they experienced the flow of time on the day of the survey.
Change in the score of Visual Analog Scale (VAS) | 2 weeks
  Subjective experience of time was measured by the VAS, which consists of a 100-mm vertical line representing the experience of time from slowest (i.e., -50 mm) to fastest (i.e., +50 mm). In this nonverbal dimensional task, subjects were asked to label how fast or slow they experienced the flow of time on the day of the survey.
Change in the score of Visual Analog Scale (VAS) | 6 weeks
  Subjective experience of time was measured by the VAS, which consists of a 100-mm vertical line representing the experience of time from slowest (i.e., -50 mm) to fastest (i.e., +50 mm). In this nonverbal dimensional task, subjects were asked to label how fast or slow they experienced the flow of time on the day of the survey.
Change in the score of Motor Agitation and Retardation Scale | Baseline
  The Motor Agitation and Retardation Scale (MARS) is designed to assess psychomotor deficits in depressed patients and consists of five major body categories including eyes, face, voice, limbs, and trunk. The severity of each item ranges from 1 to 4, with 4 being the most severe. It takes an estimated 10 to 15 minutes to complete the assessment. The descriptions and explanations of the items are intended to be simple and practical.
Change in the score of Motor Agitation and Retardation Scale | 1 week
  The Motor Agitation and Retardation Scale (MARS) is designed to assess psychomotor deficits in depressed patients and consists of five major body categories including eyes, face, voice, limbs, and trunk. The severity of each item ranges from 1 to 4, with 4 being the most severe. It takes an estimated 10 to 15 minutes to complete the assessment. The descriptions and explanations of the items are intended to be simple and practical.
Change in the score of Motor Agitation and Retardation Scale | 2 weeks
  The Motor Agitation and Retardation Scale (MARS) is designed to assess psychomotor deficits in depressed patients and consists of five major body categories including eyes, face, voice, limbs, and trunk. The severity of each item ranges from 1 to 4, with 4 being the most severe. It takes an estimated 10 to 15 minutes to complete the assessment. The descriptions and explanations of the items are intended to be simple and practical.
Change in the score of Motor Agitation and Retardation Scale | 6 weeks
  The Motor Agitation and Retardation Scale (MARS) is designed to assess psychomotor deficits in depressed patients and consists of five major body categories including eyes, face, voice, limbs, and trunk. The severity of each item ranges from 1 to 4, with 4 being the most severe. It takes an estimated 10 to 15 minutes to complete the assessment. The descriptions and explanations of the items are intended to be simple and practical.
Hamilton Depression Scale (24-items) Total Score Change | 1 weeks
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. The higher scores representing more severe levels of depression. Remission is defined as HAM-D24 ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.
Hamilton Depression Scale (24-items) Total Score Change | 6 weeks
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. The higher scores representing more severe levels of depression. Remission is defined as HAM-D24 ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.
Change in the rate of Hamilton Anxiety Scale score | Baseline
  Hamilton Anxiety Scale is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients. Each item on the scale is rated on a 5-point scale from 0 (not present) to 4 (severe), with the total score ranging from 0 to 68. Higher scores indicate higher levels of anxiety. The HAMA-17 is often used in clinical and research settings to assess the severity of anxiety symptoms and to evaluate the effectiveness of treatments for anxiety. It is a more comprehensive version of the HAMA that includes additional items to capture a broader range of anxiety symptoms.
Change in the rate of Hamilton Anxiety Scale score | 1 week
  Hamilton Anxiety Scale is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients. Each item on the scale is rated on a 5-point scale from 0 (not present) to 4 (severe), with the total score ranging from 0 to 68. Higher scores indicate higher levels of anxiety. The HAMA-17 is often used in clinical and research settings to assess the severity of anxiety symptoms and to evaluate the effectiveness of treatments for anxiety. It is a more comprehensive version of the HAMA that includes additional items to capture a broader range of anxiety symptoms.
Change in the rate of Hamilton Anxiety Scale score | 2 weeks
  Hamilton Anxiety Scale is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients. Each item on the scale is rated on a 5-point scale from 0 (not present) to 4 (severe), with the total score ranging from 0 to 68. Higher scores indicate higher levels of anxiety. The HAMA-17 is often used in clinical and research settings to assess the severity of anxiety symptoms and to evaluate the effectiveness of treatments for anxiety. It is a more comprehensive version of the HAMA that includes additional items to capture a broader range of anxiety symptoms.
Change in the rate of Hamilton Anxiety Scale score | 6 weeks
  Hamilton Anxiety Scale is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients. Each item on the scale is rated on a 5-point scale from 0 (not present) to 4 (severe), with the total score ranging from 0 to 68. Higher scores indicate higher levels of anxiety. The HAMA-17 is often used in clinical and research settings to assess the severity of anxiety symptoms and to evaluate the effectiveness of treatments for anxiety. It is a more comprehensive version of the HAMA that includes additional items to capture a broader range of anxiety symptoms.
the Chinese version of the Snaith-Hamilton Pleasure Scale | Baseline
  The Chinese version of the Snaith-Hamilton Pleasure Scale is a tool to assess pleasure deficit in depressed patients. A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score from 14 to 56. The higher the score, the more severe the pleasure deficit.
the Chinese version of the Snaith-Hamilton Pleasure Scale | 1 week
  The Chinese version of the Snaith-Hamilton Pleasure Scale is a tool to assess pleasure deficit in depressed patients. A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score from 14 to 56. The higher the score, the more severe the pleasure deficit.
the Chinese version of the Snaith-Hamilton Pleasure Scale | 2 weeks
  The Chinese version of the Snaith-Hamilton Pleasure Scale is a tool to assess pleasure deficit in depressed patients. A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score from 14 to 56. The higher the score, the more severe the pleasure deficit.
the Chinese version of the Snaith-Hamilton Pleasure Scale | 6 weeks
  The Chinese version of the Snaith-Hamilton Pleasure Scale is a tool to assess pleasure deficit in depressed patients. A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score from 14 to 56. The higher the score, the more severe the pleasure deficit.
Change in the rate of Beck Scale of Suicidal Ideation score | Baseline
  Beck Scale of Suicidal Ideation is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week. The BSI score ranges from 0 to 63, with higher scores indicating worse outcomes and lower scores indicating better outcomes.
Change in the rate of Beck Scale of Suicidal Ideation score | 1 week
  Beck Scale of Suicidal Ideation is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week. The BSI score ranges from 0 to 63, with higher scores indicating worse outcomes and lower scores indicating better outcomes.
Change in the rate of Beck Scale of Suicidal Ideation score | 2 weeks
  Beck Scale of Suicidal Ideation is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week. The BSI score ranges from 0 to 63, with higher scores indicating worse outcomes and lower scores indicating better outcomes.
Change in the rate of Beck Scale of Suicidal Ideation score | 6 weeks
  Beck Scale of Suicidal Ideation is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week. The BSI score ranges from 0 to 63, with higher scores indicating worse outcomes and lower scores indicating better outcomes.
Change in the Laukes Emotional Intensity Scale score | Baseline
  The Laukes Emotional Intensity Scale (LEIS) was one of the first instruments successfully used to assess emotional retardation due to SSRI. The scale is a self-report scale designed to evaluate a subject's emotional intensity rather than frequency. The assessment consists of 18 questions on a 5-point scale assessing the subject's emotional state compared to "usual". The total score ranges from -36 to 36, representing very low to very high emotional intensity.
Change in the Laukes Emotional Intensity Scale score | 1 week
  The Laukes Emotional Intensity Scale (LEIS) was one of the first instruments successfully used to assess emotional retardation due to SSRI. The scale is a self-report scale designed to evaluate a subject's emotional intensity rather than frequency. The assessment consists of 18 questions on a 5-point scale assessing the subject's emotional state compared to "usual". The total score ranges from -36 to 36, representing very low to very high emotional intensity.
Change in the Laukes Emotional Intensity Scale score | 2 weeks
  The Laukes Emotional Intensity Scale (LEIS) was one of the first instruments successfully used to assess emotional retardation due to SSRI. The scale is a self-report scale designed to evaluate a subject's emotional intensity rather than frequency. The assessment consists of 18 questions on a 5-point scale assessing the subject's emotional state compared to "usual". The total score ranges from -36 to 36, representing very low to very high emotional intensity.
Change in the Laukes Emotional Intensity Scale score | 6 weeks
  The Laukes Emotional Intensity Scale (LEIS) was one of the first instruments successfully used to assess emotional retardation due to SSRI. The scale is a self-report scale designed to evaluate a subject's emotional intensity rather than frequency. The assessment consists of 18 questions on a 5-point scale assessing the subject's emotional state compared to "usual". The total score ranges from -36 to 36, representing very low to very high emotional intensity.
Change in the Clinically Useful Depression Outcome Scale-Mixed Subscale score | Baseline
  The Useful Depression Outcome Scale-Mixed Subscale (CUDOS-M) is a revised scale based on the CUDOS with items added and subtracted, combining the criteria for evaluating typical manic/hypomanic episodes and depressive episodes; it is a self-assessment scale used for prognostic assessment of patients with depressive disorders with 13 rating items. Total score from 0 to 52, the higher the score the more serious the situation is.
Change in the score of THINC-it | Baseline
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it consist of 1 subjective (5-item Cognitive Impairment in Depression Questionnaire) and 4 objective (Choice Reaction Time, 1-Back Memory Task, Digit Symbol Replacement Test, and the Connectivity Test). The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in the score of THINC-it | 1 week
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it consist of 1 subjective (5-item Cognitive Impairment in Depression Questionnaire) and 4 objective (Choice Reaction Time, 1-Back Memory Task, Digit Symbol Replacement Test, and the Connectivity Test). The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in the score of THINC-it | 2 weeks
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it consist of 1 subjective (5-item Cognitive Impairment in Depression Questionnaire) and 4 objective (Choice Reaction Time, 1-Back Memory Task, Digit Symbol Replacement Test, and the Connectivity Test). The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in the score of THINC-it | 6 weeks
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it consist of 1 subjective (5-item Cognitive Impairment in Depression Questionnaire) and 4 objective (Choice Reaction Time, 1-Back Memory Task, Digit Symbol Replacement Test, and the Connectivity Test). The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in electroencephalogram | Baseline
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with TRD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of TRD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include: Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Change in electroencephalogram | 1 week
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with TRD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of TRD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include: Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Change in electroencephalogram | 2 weeks
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with TRD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of TRD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include: Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Change in electroencephalogram | 6 weeks
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with TRD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of TRD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include: Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Change in the TMS-EEG data | Baseline
  Transcranial magnetic stimulation induces changes in cortical plasticity that can persist long after the end of stimulation. EEG is the sum of excitatory and inhibitory postsynaptic potentials, reflecting the rhythmic activity of neurons in the cerebral cortex.The stimulus response characteristics of TMS-EEG can be used to measure the cortical effects induced by TMS, to explore the functions of various brain regions, to correlate the causal relationship of inter-brain interactions, as well as to diagnose and treat depression based on abnormal response characteristics.
Change in the TMS-EEG data | 1 week
  Transcranial magnetic stimulation induces changes in cortical plasticity that can persist long after the end of stimulation. EEG is the sum of excitatory and inhibitory postsynaptic potentials, reflecting the rhythmic activity of neurons in the cerebral cortex.The stimulus response characteristics of TMS-EEG can be used to measure the cortical effects induced by TMS, to explore the functions of various brain regions, to correlate the causal relationship of inter-brain interactions, as well as to diagnose and treat depression based on abnormal response characteristics.
Change in the TMS-EEG data | 2 weeks
  Transcranial magnetic stimulation induces changes in cortical plasticity that can persist long after the end of stimulation. EEG is the sum of excitatory and inhibitory postsynaptic potentials, reflecting the rhythmic activity of neurons in the cerebral cortex.The stimulus response characteristics of TMS-EEG can be used to measure the cortical effects induced by TMS, to explore the functions of various brain regions, to correlate the causal relationship of inter-brain interactions, as well as to diagnose and treat depression based on abnormal response characteristics.
IL-6 level | Baseline
  Detection of serum IL-6 levels using flow cytometry. The normal value is 0-5.30 pg/ml. There is a goodcorrelation between depression and elevated serum IL-6 levels.
IL-6 level | 1 week
  Detection of serum IL-6 levels using flow cytometry. The normal value is 0-5.30 pg/ml. There is a goodcorrelation between depression and elevated serum IL-6 levels.
IL-6 level | 2 weeks
  Detection of serum IL-6 levels using flow cytometry. The normal value is 0-5.30 pg/ml. There is a goodcorrelation between depression and elevated serum IL-6 levels.
IL-6 level | 6 weeks
  Detection of serum IL-6 levels using flow cytometry. The normal value is 0-5.30 pg/ml. There is a goodcorrelation between depression and elevated serum IL-6 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China